CLINICAL TRIAL: NCT02166411
Title: Laparoscopic Myomectomy Using Barbed or Conventional Sutures . A Randomized Controlled Trial
Brief Title: Laparoscopic Myomectomy Using Barbed or Conventional Sutures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Usama M Fouda, M.D, PhD, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: lap.myomectomy
Record Dates: First submitted 2014-06-16; First posted 2014-06-18 (Estimated); Last update posted 2020-03-13 (Actual); Status verified 2019-10

CONDITIONS: Fibroid
Keywords: Myomectomy ,Laparoscopy , Barbed sutures
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- myomectomy using barbed sutures (Experimental): .Myoma bed is sutured with barbed sutures
  Interventions: Procedure: myomectomy using barbed sutures
- myomectomy using conventional sutures (Active Comparator): Myoma bed is sutured with conventional sutures
  Interventions: Procedure: myomectomy using conventional sutures

INTERVENTIONS:
Procedure: myomectomy using barbed sutures — A transverse incision will be made over the myoma using unipolar hook and a cleavage plane between the myoma and uterus will be developed by sharp dissection. After the identification of the cleavage plane, the fibroid will be enucleated by means of adequate traction with a strong grasper and countertraction maneuvers with another grasping forceps . Bipolar forceps will be used to coagulate bleeding points . The myometrial edges will be reapproximated in one or two layers (according to the depth of the uterine wound) by using a 24-cm × 24-cm 0 polydioxanone double-armed suture on a 26-mm half-circle reverse cutting needle( STRATAFIX™ Spiral PDO Knotless Tissue Control Device, Ethicon Inc , Somerville, NJ, USA ).
  Arms: myomectomy using barbed sutures
Procedure: myomectomy using conventional sutures — A transverse incision will be made over the myoma using unipolar hook and a cleavage plane between the myoma and uterus will be developed by sharp dissection. After the identification of the cleavage plane, the fibroid will be enucleated by means of adequate traction with a strong grasper and countertraction maneuvers with another grasping forceps . Bipolar forceps will be used to coagulate bleeding points . Myometrial edges will be re-approximated using 1-0 polyglactin 910 suture(VICRYL™.; Ethicon Inc, Sommerville, NJ)
  Arms: myomectomy using conventional sutures

SUMMARY:
The aim of this study is to compare operative data and early postoperative outcomes of laparoscopic myomectomy using barbed sutures with those of laparoscopic myomectomy using conventional sutures .

DETAILED DESCRIPTION:
• Till now , there is only one small randomized controllrd study (n=22 in each arm) which compared the use of barbed suture with conventional suture in laparoscopic myomectomy .The myoma bed was closed with either conventional polyglactin suture or unidirectional barbed suture . The operative time was shorter in the barbed suture group (73.3 ± 21.4 min Vs. 80.7 ± 18.6 min) but this difference failed to reach statistical significance because of small sample size . However, the time required to suture the myoma beds was significantly lower in the barbed suture group .

ELIGIBILITY:
Inclusion Criteria:

* the presence of one to three symptomatic intramural or subserosal myomas (with largest fibroid diameter less than 10 cm).

Exclusion Criteria:

* submucosal myoma
* calcified myomas
* uterine size more than 16 weeks
* suspension of genital malignancy
* coagulation defects or concurrent anticoagulant therapy
* pregnancy
* compromised cardiopulmonary status
* previous treatment with gonadotropin-releasing hormone analogue
* contraindications for general anesthesia.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Operative time | During myomectomy operation

SECONDARY OUTCOMES:
Suturing time of myoma bed | During myomectomy operation

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Zayed, M.D,PhD, Study Chair — Cairo university ,Faculty of medicine , Obstetrics and Gynecology Department; Usama M Fouda, M.D,PhD, Study Director — Cairo university ,Faculty of medicine , Obstetrics and Gynecology Department; Khaled A Elsetohy, M.D,PhD, Principal Investigator — Cairo university ,Faculty of medicine , Obstetrics and Gynecology Department
Locations (1):
- Obstetrics &Gynecology Department , Faculty of medicine ,Cairo university, Cairo, Egypt

REFERENCES:
- [Background] Greenberg JA, Einarsson JI. The use of bidirectional barbed suture in laparoscopic myomectomy and total laparoscopic hysterectomy. J Minim Invasive Gynecol. 2008 Sep-Oct;15(5):621-3. doi: 10.1016/j.jmig.2008.06.004. Epub 2008 Jul 10. PMID 18619922